CLINICAL TRIAL: NCT02060890
Title: A Pilot Trial Testing the Feasibility of Using Molecular Profiling to Guide an Individualized Treatment Plan in Adults With Recurrent/Progressive Glioblastoma
Brief Title: Molecular Profiling in Guiding Individualized Treatment Plan in Adults With Recurrent/Progressive Glioblastoma
Acronym: TGEN
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Translational Genomics Research Institute (Other); The Ben & Catherine Ivy Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CC14101; NCI-2017-00467 (Registry Identifier: CTRP (Clinical Trial Reporting Program)
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2020-07

CONDITIONS: Adult Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surgery is done and a "core" specimen (from the enhancing component of tumor) and one or more tissue biopsies of the surrounding "rim" are obtained and processed for shipment to TGen for NGS and transcriptome profiling.
  Blood is obtained prior to and 24 hours following surgery for assessment of any circulating tumor DNA in blood.
  Blood for circulating tumor DNA is collected every 28 days (+/- 7 days).
  Whole blood samples will be immediately sent to Ashion for extraction of DNA. Isolated DNA will be quantitated by spectrophotometry, and the distribution of molecular weights in the preparations will be visualized by gel electrophoresis. Blood derived DNA samples will be aliquoted and kept at Ashion at -20 degrees Celsius until use in molecular studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Group A: Patients will undergo collection of tumor at the time of tumor resection and after confirmation of tumor progression and will have blood samples drawn pre-surgery and during standard of care follow-up visits. Patients will then be provided with a specialized tumor board recommendations for personalized treatment options for up to 4 medications based on the specimen analysis results within 35 days of surgery. Patients may then elect to initiate recommended therapy within 42 days of surgery.
  Interventions: Other: specialized tumor board recommendation

INTERVENTIONS:
Other: specialized tumor board recommendation — feasibility of a specialized tumor board to come up with treatment recommendations no later than 35 days from surgery.
  Other Names: standard of care therapy

SUMMARY:
This current study will use a new treatment approach based on each patient's tumor genomic profiling consisting of whole genome sequencing, exome analysis, and RNA sequencing as well as predictive modeling. This new treatment strategy has shown promising results in adult patients with other solid tumors.

DETAILED DESCRIPTION:
Patients with recurrent glioblastoma who are candidates for surgery for their clinical management will have tumor tissue taken at the time of surgery. Tissue samples will be obtained from the contrasting edge as well as infiltrating margins. Circulating tumor DNA will also be taken from blood samples before, and after surgery and every 2 months. Genomic profiling of the tumor tissue will be performed and a Molecular Tumor Board will review the profiling within 28 to 35 days of surgery. If specific potential targets are amenable to treatment, a treatment recommendation will be made. Up to 4 drugs could be suggested to the treating physician. The patient and the treating physician may or may not choose to use the recommendation. Any drug from the US Pharmacopeia may be chosen. If the treatment as suggested is given, patients will be followed for toxicity and efficacy, including progression and survival. If the treatment is not given, patients will be followed for progression and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand and provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization prior to initiation of any study-specific procedures
* Have a life expectancy of at least 3 months
* Patients must have a diagnosis of histologically confirmed Glioblastoma that is felt on imaging to be progressive despite standard of care treatment
* at least 18 years of age
* Patient is a good medical candidate for a standard of care surgical procedure
* Patients may enroll independent of number of prior therapies, but must have received prior radiation therapy
* Patients must have a performance status (KPS) of at least 60.

Exclusion Criteria:

* Uncontrolled concurrent illness including psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent

Eligibility for treatment using the specialized Tumor Board recommendations

* Patients must have fully recovered from any toxicity associated with surgery
* Must begin treatment no longer than 35 calendar days from surgery
* Must have KPS at least 60
* Must have Absolute Neutrophil Count (ANC) at least 1500/mm3, platelets at least 125,000/mm2, Hg at least 8 gm/dl
* Must have electrolytes (Na, K, Co2, Cl) within normal limits using institutional guidelines
* Must have baseline MRI within 14 days prior to starting cycle 1, day 1 of treatment (+/- 3 days)
* Additional laboratory guidelines will be based upon therapies suggested by the specialized Tumor Board based upon anticipated, known toxicities of those agents and must be within at least 1.5 x upper normal limits of institutional normal limits
* Patient must agree to follow the recommended treatment regimen, including clinic visits, laboratory, imaging, and toxicity assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with recurrent or progressive glioblastoma that are eligible for surgical resection.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-09-03 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Patients will undergo collection of tumor at the time of tumor resection and after confirmation of tumor progression and will have blood samples drawn pre-surgery and during standard of care follow-up visits. Patients will then be provided with a specialized tumor board recommendations for personalized treatment options for up to 4 medications based on the specimen analysis results within 35 days of surgery. Patients may then elect to initiate recommended therapy within 42 days of surgery.
  specialized tumor board recommendation: feasibility of a specialized tumor board to come up with treatment recommendations no later than 35 days from surgery.
Period: Overall Study
Arm/Group | Treatment Group
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Group A
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Treatment Recommendations Within 35 Days of Surgery
Description: To demonstrate feasibility, we would want the treatment recommendation to be fully complete within 35 calendar days in at least 85% of patients for which sufficient RNA and DNA is available.
Time Frame: 35 days from surgery to making genomic informed treatment recommendation
Population: 16 pts had tumor tissue for analysis; 15 of 16 patients received treatment recommendations within 35 days of surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A
Number analyzed (Participants) | 16
Participants | 15

2. Secondary Outcome: Number of Patients Who Chose to Pursue Treatment
Description: Number of patients who chose to pursue treatment based on these genomics-informed treatment recommendations
Time Frame: Within 35 days from surgery to making genomic informed treatment recommendation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 7

3. Other Pre Specified Outcome: Successful Generation of Patient-derived Xenograft (PDX) Genomic Models
Description: Number of patient-derived xenograft (PDX) models successfully derived from patient tumor samples.
Time Frame: Within 12 months after tissue collection
Population: Nine patients had sufficient tissue sent for PDX model development.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 9
Participants | 5

4. Other Pre Specified Outcome: Number of Participants Reaching 12 Months Progression Free Survival
Description: Treatment efficacy derived from specialized Tumor Board suggestion, defined by 12 month progression free survival.
Time Frame: 12 month progression free survival
Population: Number of patients who chose to pursue treatment based on genomic informed recommendations
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Groups:
- Group A: Patients pursuing treatment after tumor board's genomics-informed treatment recommendation.
Arm/Group | Group A
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=7)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Lung infection
seizure (Nervous system disorders) | 2 (2) — Seizure
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No